CLINICAL TRIAL: NCT02480140
Title: Self-regulated Constraint-induced Movement Therapy in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Sydney (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Karen Liu, Associate Professor, University of Western Sydney
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SR-CIMT
Record Dates: First submitted 2015-06-18; First posted 2015-06-24 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Stroke
Keywords: Self-regulation; Constraint-induced movement therapy; Stroke; Functional recovery; Randomized controlled trial
MeSH Terms: conditions — Stroke; Self-Control | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Self-regulated constraint-induced movement therapy (Experimental): Self-regulated constraint-induced movement therapy (SR-CIMT) - participants' non-hemiplegic arm was restrained in a mitt for 4 hours every day, 2 weeks, 5 days a week (therapy days) (CIMT) (the same CIMT protocol as in the CIMT group described under 'comparator/control treatment'); participants were taught using the self-regulation (SR) strategy to relearn the tasks; SR strategy involved participants self reflecting on their abilities and deficits in performing the tasks, identifying problems and solutions in achieving the most independence in the tasks, and then actually carrying out the tasks.
  Interventions: Other: Self-regulated constraint-induced movement therapy
- Constraint-induced movement therapy (Active Comparator): In the constraint-induced movement therapy group (CIMT), participants' non-hemiplegic arm was restrained in a mitt for 4 hours every day, 2 weeks, 5 days a week (therapy days); therapist provided demonstration on the adapted task performance with one arm (the side of participants' hemiplegic arm), and participants to practice the tasks with the unrestrained hemiplegic arm under supervision.
  Interventions: Other: Constraint-induced movement therapy
- Conventional occupational therapy (Active Comparator): It involved therapist to demonstrate the adapted task performance followed by patient's practice under supervision.
  Interventions: Other: Conventional occupational therapy

INTERVENTIONS:
Other: Self-regulated constraint-induced movement therapy — There were 10 tasks to practice in total, they included fold laundry, put clothes on hanger, brush teeth, dress upper garment, dress lower garment in week one; and use telephone, prepare a cup of tea, sweep floor, wash towel, wash dishes in week two. In the 4 hours when the participants had their non-hemiplegic arm in the restrain, they received one hour therapist-guided training using SR strategy on task relearning as described above. Therefore, all participants received 10 one-hour therapist-guided training sessions (daily on weekdays, total two weeks). The intervention was delivered by occupational therapist. For the rest of the 3 hours in the restrain, the participants' wearing of the restrain was monitored by the nursing staff in the ward.
  Arms: Self-regulated constraint-induced movement therapy
Other: Constraint-induced movement therapy — They practised the same 10 tasks as in the SR-CIMT and control groups. The same as the experimental intervention group (SR-CIMT), in the 4 hours when the participants had their non-hemiplegic arm in the restrain, they received one hour therapist-guided training using the strategy on task relearning as described above. Therefore, all participants received 10 one-hour therapist-guided training sessions (daily on weekdays, total two weeks). The intervention was delivered by occupational therapist. For the rest of the 3 hours in the restrain, the participants' wearing of the restrain was monitored by the nursing staff in the ward.
  Arms: Constraint-induced movement therapy
Other: Conventional occupational therapy — They practised the same 10 tasks as in the SR-CIMT group described above. They received training for 2 weeks, 5 days a week (therapy days), the same as in the SR-CIMT and CIMT groups.
  Arms: Conventional occupational therapy

SUMMARY:
Emerging research suggests the use of self-regulation (SR) strategies at improving functional regain in patients with brain injury. SR is proposed to produce an added effect to the effective constraint-induced movement therapy (CIMT). This study aimed to examine the efficacy of a self-regulated CIMT program (SR-CIMT) for function regain of patients with subacute stroke. It was hypothesized that participants receiving the combined treatment (SR and CIMT) would have a better functional regain.

DETAILED DESCRIPTION:
Background - Emerging research suggests the use of self-regulation (SR) strategies at improving functional regain in patients with brain injury. SR is proposed to produce an added effect to the effective constraint-induced movement therapy (CIMT).

Objective - This study aimed to examine the efficacy of a self-regulated CIMT program (SR-CIMT) for function regain of patients with sub-acute stroke.

Methods - Seventy-six patients were randomly assigned to the self-regulated constraint-induced movement therapy (SR-CIMT; n=25), constraint-induced movement therapy (CIMT; n=27) or conventional functional rehabilitation (control; n=24) groups, and completed the trial.

The SR-CIMT intervention was two-week therapist-guided training using the SR strategy to reflect on the relearning of functional tasks with CIMT. Outcome measurements were for upper limb function (Action Research Arm Test, ARAT, Fugl-Meyer Assessment, FMA), daily task performance (Lawton Instrumental Activities of Daily Living Scale, Lawton IADL) and self-perceived functional ability (Motor Activity Log, MAL) at pre and post intervention intervals, and at one month follow up.

ELIGIBILITY:
Inclusion Criteria:

* sustained an ischemic type stroke with lesion in the primary or motor cortical areas resulting in hemiplegia,
* had stroke onset of less than 3 months,
* were aged above 60, and
* had 10 degree active extension in metacarpophalangeal joint and interphalangeal joint, 20 degree active extension of wrist joint

Exclusion Criteria:

* had excessive spasticity in the affected limb, as defined by a score of 2 or more on the Modified Ashworth Scale,
* had excessive pain in the affected limb, as defined by a score 4 or more using a Visual Analog Scale,
* had a score below 19 on the Mini-Mental Status Examination (MMSE), and
* had diagnosed of depression according to Diagnostic and Statistical Manual-IV (DSM-IV) criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Lawton Instrumental Activities of Daily Living Scale after the intervention | Baseline and after the intervention (2 weeks)
  Performance assessment on 8 daily tasks
Change from baseline in Lawton Instrumental Activities of Daily Living Scale at one month after the intervention completed | Baseline and one month after the intervention completed (1 month and 2 weeks)
  Performance assessment on 8 daily tasks
Change from baseline in Action Research Arm Test after the intervention | Baseline and after the intervention (2 weeks)
  Performance assessment on arm function
Change from baseline in Action Research Arm Test at one month after the intervention completed | Baseline and one month after the intervention completed (1 month and 2 weeks)
  Performance assessment on arm function
Change from baseline in Fugl Meyer Assessment, upper extremity motor subsection after the intervention | Baseline and after the intervention (2 weeks)
  Performance assessment on arm function
Change from baseline in Fugl Meyer Assessment, upper extremity motor subsection at one month after the intervention completed | Baseline and one month after the intervention completed (1 month and 2 weeks)
  Performance assessment on arm function

SECONDARY OUTCOMES:
Change from baseline in Motor Activity Log-28 after the intervention | Baseline and after the intervention (2 weeks)
  Self-reported assessment on daily function
Change from baseline in Motor Activity Log-28 at one month after the intervention completed | Baseline and one month after the intervention completed (1 month and 2 weeks)
  Self-reported assessment on daily function

CONTACTS AND LOCATIONS:
Overall Officials: Karen P.Y. Liu, PhD, Principal Investigator — University of Western Sydney
Locations (2):
- Hong Kong (2):
  - Shatin Hospital, Hong Kong
  - Pok Oi Hospital, Yuen Long

REFERENCES:
- [Background] Lam, K., Liu, K., Leung, T., Sum, C., Yue, A. & Mok, V. (2013, 24-26 July). The effectiveness of self-regulated constraint-induced movement therapy for functional regain for people with sub-acute stroke: A randomized controlled trial. Australian Occupational Therapy Journal, 110.
- [Background] Leung, T., Liu, K.P.Y., Sum, C., Mok, V. & Lum, C. (2010). Self-regulation constraint-induced movement therapy programme for people with subacute stroke. Hong Kong Hospital Authority Rehabilitation Symposium.
- [Background] Leung, T., Liu, K.P.Y., Sum, C., Mok, V. & Lum, C. (2010). Self-regulation constraint-induced movement therapy programme for people with subacute stroke. Hong Kong Journal of Occupational Therapy,19, A8.